CLINICAL TRIAL: NCT04981197
Title: Effects of Baduanjin Exercise on Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13-S-013
Record Dates: First submitted 2021-07-18; First posted 2021-07-28 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
Keywords: heart failure; Baduanjin exercise; fatigue; sleep quality; psychological distress; quality of life
MeSH Terms: conditions — Heart Failure; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin exercise group (Experimental): The Baduanjin exercise group received a 12-week Baduanjin exercise programme.
  Interventions: Behavioral: Baduanjin exercise
- Control group (No Intervention): Patients in this group maintain their daily life activities, and there is no intervention given.

INTERVENTIONS:
Behavioral: Baduanjin exercise — Patients in the intervention group underwent a 12-week Baduanjin exercise programme consisting of 12 weeks of Baduanjin exercise, a 35-min Baduanjin exercise demonstration video, a picture-based educational brochure, and a performance record form.
  Arms: Baduanjin exercise group

SUMMARY:
This study was a parallel, randomized controlled trial with a longitudinal research design. Participants were randomly assigned to either the Baduanjin exercise group or the control group. The Baduanjin exercise group received a 12-week Baduanjin exercise programme. The control group received usual care. Fatigue, sleep quality, psychological distress, quality of life were assessed by a structured questionnaire at baseline, 4 weeks, 8 weeks, and 12 weeks after enrollment.

DETAILED DESCRIPTION:
This study was a parallel, randomized controlled trial with a longitudinal research design. Participants were randomly assigned to either the Baduanjin exercise group or the control group. Patients in the intervention group underwent a 12-week Baduanjin exercise programme consisting of 12 weeks of Baduanjin exercise, a 35-min Baduanjin exercise demonstration video, a picture-based educational brochure, and a performance record form. The control group received usual care. Fatigue, sleep quality, psychological distress, quality of life were assessed by a structured questionnaire at baseline, 4 weeks, 8 weeks, and 12 weeks after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stable heart failure by a physician according to the New York Heart Association (NYHA) class I and II
* Aged 20 years or older
* Able to communicate and speak Chinese
* Have video devices available to use at home

Exclusion Criteria:

* Impaired mobility, defined as a limitation in independent, purposeful physical movement of the body or of one or more extremities
* Unstable angina or myocardial infarction, unstable serious arrhythmia, unstable structural valvular disease, open-heart surgery, or chronic obstructive pulmonary disease (COPD)
* Diagnosis of major depression and cognitive disorders
* Unstable vital signs (defined as blood pressure > 180/110 mmHg or < 90/60 mmHg and resting heart rate > 100 beats/min).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-12-17 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in the modified Piper Fatigue Scale scores | baseline, 4 week, 8 week, 12 week
  Changes from baseline modified Piper Fatigue scale at 4 weeks, 8 weeks, 12 weeks.The shortened modified Piper Fatigue scale is composed of 15 items that measure two domains of fatigue: severity and temporality. Each item is scored from 0 to 3, with a total possible score of 0-45. Higher scores indicate greater fatigue.
Changes in the Minnesota Living with Heart Failure Questionnaire scores | baseline, 4 week, 8 week, 12 week
  Changes from baseline Minnesota Living with Heart Failure Questionnaire at 4 weeks, 8 weeks, 12 weeks.The Minnesota Living with Heart Failure Questionnaire is composed of 21 items. Each item score ranges from 0 to 5. The total possible score ranges from 0 to 105, with higher scores indicating a lower quality of life.

SECONDARY OUTCOMES:
Changes in the Pittsburgh Sleep Quality Index scores | baseline, 4 week, 8 week, 12 week
  Changes from baseline Pittsburgh Sleep Quality Index at 4 weeks, 8 weeks, 12 weeks.The Pittsburgh Sleep Quality Index is composed of 21 items, 7 dimensions. Each dimension is scored from 0 to 3, with a total possible score of 0-21. Higher scores indicate poor sleep.
Changes in the Hospital Anxiety and Depression Scale scores | baseline, 4 week, 8 week, 12 week
  Changes from baseline Hospital Anxiety and Depression Scale at 4 weeks, 8 weeks, 12 weeks.The Hospital Anxiety and Depression Scale is composed of 14 items, 2 subscales. Each item is scored from 0 to 3, with a total possible score of 0-21 for each subscale. Higher scores indicate higher anxiety and depression
Changes in heart rate variability | baseline, 4 week, 8 week, 12 week
  Changes from baseline heart rate variability at 4 weeks, 8 weeks, 12 weeks.The heart rate variability was measured using the "Heart Rate Master ANSWatch® Wrist Physiological Monitor TS-0411Deluxe Advanced" (made in Taiwan)

IPD SHARING:
Plan to Share IPD: No